CLINICAL TRIAL: NCT05950815
Title: A Phase I Study to Evaluate the Tolerance, Safety, Pharmacokinetic Characteristics and Preliminary Efficacy of PM1015 in Patients With Advanced Solid Tumors
Brief Title: A Study of PM1015 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PM1015-A001M-ST-R
Record Dates: First submitted 2023-05-18; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — 5'-Nucleotidase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM1015 (Experimental): Subjects will be administered PM1015 via intravenously (IV) once in first cycle, then administered PM1015 every 2 weeks (Q2W ) after 3 weeks
  Interventions: Drug: CD73 Antigen

INTERVENTIONS:
Drug: CD73 Antigen — subjects will be administered with PM1015 via intravenously (IV) Q2W pemetrexed until progression or accepted other treatment.
  Other Names: PM1015 injection

SUMMARY:
PM1015 is a specific antibody targeting CD73. This is a phase I study to evaluate the efficacy and safety of PM1015 in patients with advanced solid tumor.

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase I study contains dose escalation stage and dose expansion stage. The dose escalation stage will be following the accelerated titration design and the classic 3+3 design, with a planned enrollment of 13 to 24 patients with advanced tumors. The dose expansion stage will be used safe and tolerable doses, with a planned enrollment of 24 patients with advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in clinical trials; Fully understand the test and voluntarily sign the informed consent; Willing to follow and able to complete all test procedures;
* No gender limit, aged between 18 and 75 years (including boundary values);
* Subjects with histologically or cytologically confirmed advanced malignant solid tumors who have failed standard treatment, have no standard treatment options, or are not currently eligible for standard treatment;
* Adequate organ function, as defined below:

  1. Blood system (in the absence of blood transfusion, granulocyte colony stimulating factor, or other medical support within 14 days prior to initiation of trial therapy) : neutrophil count (ANC) >= 1.5 x 10^9 /L; Platelet count (PLT) >= 100 x 10^9 /L; Hemoglobin (Hb) >= 90 g/L;
  2. Liver function: total bilirubin (TBIL) <= 1.5 x upper limit of normal (ULN), subjects with liver metastasis or liver cancer <= 2 x ULN; Subjects with Gilbert disease should be <= 3 x ULN; Aspartate aminotransferase (AST), alanine aminotransferase (ALT) <= 2.5 x ULN (subjects with liver metastasis or liver cancer: <= 3 x ULN);
  3. Renal function: serum creatinine <= 1.5 x ULN or creatinine clearance >= 50 mL/min (Cockcroft-Gault formula: [(140 - age) x body weight (kg) x 0.85 (for females only)] / [72 x creatinine (mg/dL)]; (Creatinine unit conversion: 1 mg/dL = 88.4 μmol/L); Qualitative urine protein <= 1+; If the qualitative urine protein >= 2+, 24h urine protein quantitative examination is required; if the quantitative urine protein < 1g, it is acceptable;
  4. Coagulation function: International standardized ratio (INR) and activated partial thrombin time (APTT) should be less than 1.5 x ULN; Subjects with liver metastasis or liver cancer should be <= 2 x ULN;
* Physical status: The Eastern Cooperative Oncology Group (ECOG) physical status score was 0-1;
* Expected survival >= 12 weeks;
* Dose escalation test: According to RECIST version 1.1, there is at least one evaluable tumor lesion; Initial dose extension test: At least one measurable tumor lesion according to RECIST version 1.1; (Tumor lesions located in the area of previous radiotherapy or other local regional treatment sites are generally not considered as measurable lesions, unless the lesions show definite progression or persist 3 months after radiotherapy; Not accept only bone metastases or only central nervous system metastases as measurable lesions);
* All subjects should undergo a fresh tumor lesion biopsy during the screening period (No bone biopsy; Biopsy is also not acceptable in subjects with a single target lesion for biopsy); If biopsy is not possible, subjects should provide formalin-fixed-paraffin-embedded (FFPE) tumor samples from the nearest (up to 24 months) to the start of the trial for biomarker analysis; If the subject is unable to provide specimens that meet the above requirements due to special reasons, the subject may participate in screening with the consent of the sponsor's medical monitor;
* A fertile female subject has a negative serum-pregnancy result within 7 days prior to the start of the trial treatment and is willing to abstain from sex or use a medically approved highly effective contraceptive method (e.g. IUD, condom) from the date of signing the informed consent to 6 months after the end of the final medication;
* Male subjects are willing to abstain from sex or use a medically approved highly effective contraceptive method for 6 months from the date of signing the informed consent, and do not donate sperm during this period.

Exclusion Criteria:

* History of severe allergic disease, allergy to serious drugs (including unmarketed test drugs) or known allergy to any component of the test drug;
* Previous treatment with adenosine inhibitors (such as anti-CD73, anti-CD39, or anti-A2aR);
* Received an unmarketed investigational drug or treatment within 4 weeks prior to initiation of the trial treatment, or is still within the drug's 5 half-lives (if known), whichever is longer;
* The adverse reactions of previous antitumor therapy have not recovered to the NCI-CTCAE V5.0 rating <= grade 1 (except for toxicities without safety risks as determined by the researchers, such as hair loss, grade 2 peripheral neurotoxicity, stable hypothyroidism after hormone replacement therapy, etc.);
* Received the following treatments or drugs before starting the trial therapy:

  1. Major organ surgery (excluding needle biopsy) or major trauma or invasive dental procedures within 4 weeks before the initiation of trial treatment, or the need for elective surgery during the trial;
  2. Within 4 weeks prior to initiation of trial therapy, received chemotherapy, radical/extensive radiotherapy, endocrine therapy, biological therapy (such as tumor vaccine, cytokine), immune checkpoint agonists (such as 4-1BB agonists, OX40 agonists) or immune checkpoint inhibitors (such as anti-PD-1, anti-PD-L1, anti-CTLA-4, anti-LAG-3) and other anti-tumor therapy; Received nitrosourea and mitomycin C within 6 weeks prior to initiation of treatment; Received oral fluorouracil, small-molecule targeted drugs, and traditional Chinese medicine with anti-tumor indications within 2 weeks before the start of the experimental treatment; Received palliative radiotherapy for vital organs (such as liver, brain, lung, etc.) within 7 days prior to the start of trial therapy;
  3. Received systemic glucocorticoid (prednisone >10 mg/ day or equivalent dose of the same drug) or other immunosuppressant therapy within 14 days prior to the initial use of the test drug; Except in the following cases: treatment with topical, ocular, intra-articular, intranasal, and inhaled corticosteroids; Short-term use of glucocorticoids for preventive treatment (e.g. to prevent hypersensitivity to contrast media);
  4. Have received live attenuated vaccine within 4 weeks before the first use of the trial drug;
* History of immune deficiency, including HIV antibody positive test;
* Syphilis antibody positive;
* HBsAg or HBcAb positive, HBV-DNA > 500 IU/mL or lower limit of detection in test center (only when lower limit of detection in test center is higher than 500 IU/mL); HCV antibody positive and HCV-RNA higher than the lower limit of test center detection; 9. Subjects with brain parenchymal metastasis or meningeal metastasis with clinical symptoms were judged by the researchers to be unsuitable for inclusion;
* Active infection;
* Subjects with active or previous autoimmune diseases with potential recurrence (e.g. systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except clinically stable autoimmune thyroid disease and type I diabetes;
* Currently with uncontrollable pleural, pericardial and abdominal effusion;
* A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

  1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, degree Ⅱ-Ⅲ atrioventricular block;
  2. The mean QT interval (QTcF) corrected by Fridericia was >450 ms for male and > 470 ms for female;
  3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before trial administration began;
  4. New York Heart Association Cardiac Function Grade >= II, or left ventricular ejection fraction (LVEF) < 50%;
  5. Clinically uncontrolled hypertension (systolic blood pressure >= 160 mmHg and/or diastolic blood pressure >=100 mmHg);
  6. The presence of any factors that increase the risk of prolonged QTc or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, or the use of any concomitant drugs known to prolong the QT interval;
* Previous history of allogeneic organ transplantation or allohematopoietic stem cell transplantation;
* A known history of alcohol abuse, psychotropic substance abuse or drug use;
* Subjects with mental disorders or poor compliance;
* Pregnant or lactating subjects;
* According to the investigator's judgment, the basic condition of the subject may increase the risk of receiving the trial drug treatment, or cause confusion in the interpretation of toxic reactions and AEs;
* Other circumstances in which the investigator did not consider participation in the trial appropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | up to 21 days
  Occurrence of DLT after receiving PM1009 injection
Treatment-related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months
  Defined as the number of patients with best overall response of confirmed CR or PR per RECIST 1.1 divided by the patients with at least one tumour imaging evaluation
Disease control rate (DCR) | Up to 24 months
  Defined as the percentage of patients who have achieved CR, PR, Non-CR/Non-PD, or SD in the study.
Progression-free survival (PFS) | Up to 24 months
  Defined as the time from the date of first dose of study drug to the first observation of documented disease progression per RECIST 1.1 as determined by the Investigators or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 24 months
  Defined as the time from the date of first dose of study drug to the date of documented death due to any cause.
Anti-drug antibody (ADA) | Up to 30 days after last treatment
  PM1015 anti-drug antibody
Recommended Phase II Dose (RP2D) | Up to 30 days after last treatment
  To determine the RP2D of PM1015 injection
Maximum observed concentration (Cmax) | Up to 30 days after last treatment
  To evaluate the Cmax of PM1015 monotherapy
Time to Cmax (Tmax) | Up to 30 days after last treatment
  To evaluate the Tmax of PM1015 monotherapy
Minimum observed concentration (Cmin) | Up to 30 days after last treatment
  To evaluate the Cmin of PM1015 monotherapy
Trough concentrations (Ctrough) | Up to 30 days after last treatment
  To evaluate the Ctrough of PM1015 monotherapy
Area under the concentration-time curve (AUC0-last) | Up to 30 days after last treatment
  To evaluate the AUC0-tau of PM1015 monotherapy
Apparent terminal elimination half-life (t1/2) | Up to 30 days after last treatment
  To evaluate the t1/2 of PM1015 monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract, articles or papers) or any presentations.
Time Frame: After the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.